CLINICAL TRIAL: NCT05155709
Title: A Phase Ib/II Open Label Dose Confirmation, Proof of Concept Study of Siremadlin in Combination With Venetoclax Plus Azacitidine in Unfit Adult AML Participants Who Responded Sub-optimally to First-line Venetoclax Plus Azacitidine Treatment and in Participants With Newly Diagnosed Unfit AML Presenting With High-risk Clinical Features
Brief Title: A Study of Siremadlin in Combination With Venetoclax Plus Azacitidine in Adult Participants With Acute Myeloid Leukemia (AML) Who Are Ineligible for Chemotherapy.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After enrolling 14 patients, Novartis decided to permanently halt enrollment and terminate the siremadlin program. Consequently, enrollment for Part 2 did not commence. This decision was not influenced by any safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHDM201I12201; 2021-001165-21 (EudraCT Number)
Record Dates: First submitted 2021-10-20; First posted 2021-12-14 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; AML; Azacitidine; venetoclax; TP53; MDM2; siremadlin; HDM201; unfit adult AML participants; newly diagnosed unfit AML; presenting with high-risk clinical features
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — siremadlin; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Unfit adult participants with AML who responded sub-optimally to standard of care (Experimental): Unfit adult participants with AML who responded sub-optimally to at least 2 and not more than 4 cycles ( 1 cycle=28 days) of first-line venetoclax plus azacitidine therapy
  Interventions: Drug: siremadlin; Drug: venetoclax; Drug: azacitidine
- Arm 2: Newly diagnosed unfit adult participants with high-risk AML (Experimental): Unfit adult participants with newly diagnosed AML and with adverse genetic risk stratification (according to ELN 2022)(Except TP53 mutation positive participants).
  Interventions: Drug: siremadlin; Drug: venetoclax; Drug: azacitidine

INTERVENTIONS:
Drug: siremadlin — Siremadlin is a capsule taken orally once a day (QD) and comes in 10 mg, 20 mg and 30 mg strengths
  Other Names: HDM201
Drug: venetoclax — Venetoclax is a tablet taken orally once a day (QD) and comes in 10 mg, 50 mg and 100 mg strengths.
Drug: azacitidine — Azacitidine is a powder for suspension for injection or powder for solution for infusion taken intravenously or subcutaneously according to standard local clinical practice

SUMMARY:
A study of siremadlin in combination with venetoclax plus azacitidine in adult participants with AML who are ineligible for chemotherapy.

The primary purpose of this study was to assess whether siremadlin in combination with venetoclax plus azacitidine can enhance the clinical response in unfit AML patients without unacceptable levels of treatment-emergent toxicities.

DETAILED DESCRIPTION:
The recommended dose of siremadlin in combination with venetoclax plus azacitidine will be determined to be explored further in the expansion phase and the preliminary efficacy in achieving Complete Remission (CR) will be evaluated in participants who responded sub-optimally to first-line venetoclax plus azacitidine treatment.

The study was planned to be conducted in two parts. The primary purpose of Part 1 (Safety Run- in) was to rule out excessive toxicity of siremadlin when administered in combination with venetoclax plus azacitidine while the primary purpose of Part 2 (Expansion) was to evaluate the preliminary efficacy of siremadlin when combined with venetoclax plus azacitidine in the respective patient population.

The study treatment (siremadlin in combination with venetoclax plus azacitidine) is administered in cycles with a planned duration of 28 days and will continue until the participants experience disease progression/relapse or unacceptable toxicity.

The initial enrollment plan and safety review was as follow:

* In the Safety run-in part, 9-15 participants were planned to be enrolled in each arm. Approximately 3-6 participants were planned to be enrolled at the starting dose level of siremadlin in combination with venetoclax plus azacitidine in both arms independently. Provided the starting dose level is determined to be safe, approximately 6-9 additional participants were planned to be enrolled at dose level +1. Safety review meetings were planned to take place involving participating investigators and the Sponsor Team to make decisions regarding siremadlin dose and determine the recommended dose for expansion.
* Approximately 26 patients were planned to be treated at the recommended dose in the expansion part.

In the safety run-(Part 1) 27 sites were open for recruitment with 28 patients screened and 14 patients enrolled.

After enrolling 14 patients (6 patients in Arm 1 and 8 patients in Arm 2), Novartis took the decision to put the enrollment in permanent halt and terminate the siremadlin program. For that reason, the enrollment in Part 2 (expansion phase) will not be open. The Novartis decision was not driven by any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

- Age at the date of signing the informed consent form (ICF): Arm 1 and Arm 2: ≥ 18 years

- Participants diagnosed with AML based on WHO 2016 classification (Arber et al 2016) who are ineligible for standard induction chemotherapy and: Arm 1 : have received at least 2 cycles and not more than 4 cycles of first-line venetoclax plus azacitidine treatment and have not achieved a CR, CRi, CRh or MLFS.

Arm 2 : newly diagnosed AML with adverse genetic risk stratification (according to ELN 2022) (except TP53 mutation positive participants).

* Participant (in both arms) must be considered ineligible for standard of care intensive induction chemotherapy defined by the following:

  * 75 years of age; OR
  * 18 to 74 years of age with at least one of the following co-morbidities: Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 or 3; Cardiac history of congestive heart failure (CHF) requiring treatment or Ejection Fraction ≤ 50% or chronic stable angina; DLCO ≤ 65% or FEV1 ≤ 65%.
* Participants must have an ECOG performance status:

  0 to 2 for participants ≥ 75 years of age. OR 0 to 3 for participants ≥ 18 to 74 years of age.
* WBC < 25x109/L
* AST and ALT ≤ 3 × ULN
* Estimated Glomerular Filtration Rate (eGFR)≥ 60 mL/min/1.73 m2

Exclusion Criteria:

* Prior exposure to MDM2-inhibitor therapy at any time.
* Participants with TP53 mutation positive.
* Participants with del17p.
* Participants with AML-M3 / APL (Acute promyelocytic leukemia) with PML-RARA (Promyelocytic leukemia/retinoic acid receptor alpha) or with AML secondary to Down's syndrome.
* Participants treated with FLT3 inhibitors for AML indication are not eligible.
* Participants who require treatment with moderate or strong CYP3A4 inducers within 14 days prior to starting study treatment, or are expected to receive moderate or strong CYP3A4 inducers during the entire study
* Participants who require treatment with substrates of CYP3A4/5 with a narrow therapeutic index.

Other protocol-defined inclusion/exclusion criteria may apply at the end

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Dose Limiting Toxicities (DLTs) as per investigator assessment reported during the first cycle (separately in Arm 1 & Arm 2) | From Cycle 1 Day 1 to Cycle 1 Day 28 (28 days)
  The objective for the safety run-in is to determine the recommended dose of siremadlin in combination with venetoclax plus azacitidine to be explored further in the expansion part separately in Arm 1 and Arm 2.
Percentage of participants treated at the recommended dose for expansion, achieving a complete remission (CR) as per investigator assessment (Arm 1 only) | At least 7 cycles (196 days)
  The objective is to evaluate preliminary efficacy of siremadlin at the determined recommended dose for expansion (RDE) when administered in combination with venetoclax and azacitidine.
  This endpoint will not be analyzed since the recommended dose was not determined due to early termination.

SECONDARY OUTCOMES:
Percentage of participants treated at the recommended dose for expansion, achieving CR as per investigator assessment (Arm 2 only; for Arm 1 assessment of CR is a primary outcome measure)) | up to 3 years
  Assessment of CR in order to evaluate preliminary efficacy of siremadlin (in combination of venetoclax plus azacitidine) at the determined recommended dose for Arm 2 participants.
  This endpoint will not be analyzed since the recommended dose was not determined due to early termination.
Time of the date of the first documented CR to the date of the first documented relapse or death due to any cause, whichever occurs first (Arm 1 and Arm 2 separately) | up to 3 years
  Assessment of duration of CR in participants who achieved a CR.
  This endpoint will not be analyzed since the recommended dose was not determined due to early termination.
Percentage of participants achieving CR or complete remission with partial hematological recovery (CRh) and percentage of participants achieving CR or complete remission with incomplete hematological recovery (CRi) (Arm 1 and Arm 2) | up to 3 years
  Assessment of CR/CRh rate and CR/CRi rate.
Time from the date of the first documented CR/CRh and CR/CRi to the date of first documented relapse or death due to any cause, whichever occurs first (Arm 1 and Arm 2 separately) | up to 3 years
  Assessment of duration of CR/CRh and duration of CR/CRi.
  This endpoint will not be analyzed since the recommended dose was not determined due to early termination.
The time from start of treatment to death due to any cause (Arm 1 and Arm 2 separately) | up to 3 years
  Assessment of Overall Survival (OS).
  This endpoint will not be analyzed since the recommended dose was not determined due to early termination.
Percentage of participants died due to any cause from start of treatment until 30- and 60-day (Arm 1 and Arm 2) | 30 days & 60 days from start of study treatment
  To assess rate of early mortality at 30 day and 60 days from start of study treatment
Pharmacokinetic (PK) parameters: AUCs of siremadlin, venetoclax and azacitidine (Arm 1 and Arm 2) | up to 3 years
  AUC0-t: The area under the concentration vs. time Curve (AUC) from time zero to specified time point.
  AUClast is the AUC from time zero to the last quantifiable concentration point (last) (mass x time x volume -1).
  AUCtau is the AUC to the end of the dosing interval as when possible PK samples will be collected up to 24 h postdose for siremadlin and venetoclax. Steady-state will be assumed on Day 5 (AUCtau, ss) in case of continuous dosing.
PK parameter: Cmax of siremadlin, venetoclax and azacitidine (Arm 1 and Arm 2) | up to 3 years
  To characterize the PK of siremadlin, venetoclax and azacitidine administered in combination in each arm. Cmax is the maximum (peak) observed plasma, blood, serum or other body fluid drug concentration following drug administration (mass x volume -1)
PK parameter: Tmax of siremadlin, venetoclax and azacitidine (Arm 1 and Arm 2) | up to 3 years
  PK parameter Tmax and concentration vs time profiles of siremadlin, venetoclax and azacitidine. Tmax is the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after drug administration (time).
Percentage of CR- Measurable Residual Disease (MRD) negative overall and in participants achieving a CR, CR/CRh, and CR/CRi (Arm 1 and Arm 2) | up to 3 years
  To assess the effect of siremadlin in combination with venetoclax plus azacitidine in MRD

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (2):
  - Oregon Health Sciences University, Portland, Oregon
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Budapest, Hungary
- Israel (2):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Jerusalem
- Novartis Investigative Site, Bologna, BO, Italy
- Malaysia (2):
  - Novartis Investigative Site, Alor Star, Kedah
  - Novartis Investigative Site, Kuala Selangor
- Novartis Investigative Site, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: Novartis Results Database (NovCTRD) — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18296
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2575